CLINICAL TRIAL: NCT01609010
Title: Rituximab (Mabthera®) as Single Agent and in Combination With Interferon Alfa-2a (Roferon-A®), a Phase-III Randomized Trial in Patients With Follicular or Other CD20+ Low-grade (Indolent) Lymphoma
Brief Title: A Study of MabThera/Rituxan (Rituximab) Alone and in Combination With Roferon-A in Patients With Follicular or Other CD20+ Low-Grade (Indolent) Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML16865
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Interferon alpha-2

ARMS (2):
- Rituximab Monotherapy (Active Comparator): Participants received 375 milligrams per square meter (mg/m2) rituximab intravenously (i.v.) weekly for 4 weeks. Participants achieving minor response (MR), partial response (PR), or completer response (CR) received a second cycle of treatment.
  Interventions: Drug: rituximab
- Rituximab, Interferon (Experimental): Participants received 375 mg/m2 rituximab i.v. weekly for 4 weeks; and 3 million international units per day (MIU/day) interferon-a2a subcutaneously (s.c.) during Week 1, and 4.5 MIU/day s.c. 6 days per week during Weeks 2 through 5. Interferon-a2a was not administered on days of rituximab administration. Participants achieving MR, PR, or CR received a second cycle of treatment.
  Interventions: Drug: rituximab; Drug: interferon-a-2a

INTERVENTIONS:
Drug: rituximab — 375 mg/m2 rituximab i.v. weekly for 4 weeks
  Other Names: MabThera; Rituxan
Drug: interferon-a-2a — 3 MIU/day interferon-a2a s.c. during Week 1, and 4.5 MIU/day s.c. 6 days per week during Weeks 2 through 5
  Other Names: Roferon-A
  Arms: Rituximab, Interferon

SUMMARY:
This randomized, open-label study will compare the efficacy and safety of MabThera/Rituxan (rituximab) alone, and in combination with Roferon-A (interferon alfa-2a) in patients with follicular or other CD20+ low-grade lymphoma. Patients will be randomized to receive either MabThera/Rituxan 375 mg/m2 intravenously weekly for 4 weeks or Roferon-A 3 MIU/day subcutaneously in Week 1 followed by 4.5 MIU/day sc in Weeks 2-5 plus MabThera/Rituxan 375 mg/m2 weekly iv in Weeks 3-6. Patients who have a response will receive an additional cycle of treatment. The anticipated time on study treatment is up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years of age
* CD20+ low-grade (indolent) lymphoma of follicular and marginal zone type, small lymphocytic lymphoma without a B-CLL phenotype, or indolent lymphoma not otherwise specified
* Stage II (with bulky disease), III, or IV lymphoma
* No previous chemotherapy or a maximum of 6 months chlorambucil or cyclophosphamide
* Indication for treatment: symptomatic enlarged lymph nodes, spleen or other lymphoma manifestations, progression >6 months of lymphadenopathy or splenomegaly, anemia or thrombocytopenia or decreased hemoglobin or platelets due to lymphoma, general symptoms (weight loss, night sweats or fever)
* WHO performance status 0-2

Exclusion Criteria:

* Prior treatment with rituximab or an interferon
* B-CLL, mantle cell lymphoma, lymphoplasmacytic lymphoma (Waldenstroem's disease), or central nervous system lymphoma
* Indolent lymphoma transformed into aggressive lymphoma
* Indolent lymphoma with bulky tumor requiring urgent therapy
* Prior malignancies, except non-melanoma skin tumors, in situ cervical cancer, or curative surgery >5 years ago
* Positive for HIV infection
* Uncontrolled asthma or allergy requiring corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2002-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (29):
- Denmark (3):
  - Copenhagen
  - Hillerød
  - Roskilde
- Norway (5):
  - Bergen
  - Oslo
  - Stavanger
  - Tromsø
  - Trondheim
- Sweden (21):
  - Eskilstuna
  - Falun
  - Gothenburg
  - Halmstad
  - Huddinge
  - Jönköping
  - Karlstad
  - Kristianstad
  - Linköping
  - Luleå
  - Lund
  - Malmo
  - Örebro
  - Stockholm
  - Sundsvall
  - Uddevalla
  - Umeå
  - Uppsala
  - Vaxjo
  - Västerås
  - Visby

REFERENCES:
- [Derived] Kimby E, Ostenstad B, Brown P, Hagberg H, Erlanson M, Holte H, Linden O, Johansson AS, Ahlgren T, Wader K, Wahlin BE, Delabie J, Sundstrom C; Nordic Lymphoma Group (NLG). Two courses of four weekly infusions of rituximab with or without interferon-alpha2a: final results from a randomized phase III study in symptomatic indolent B-cell lymphomas. Leuk Lymphoma. 2015;56(9):2598-607. doi: 10.3109/10428194.2015.1014363. Epub 2015 Mar 11. PMID 25686644

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Monotherapy: Participants rituximab received 375 milligrams per square meter (mg/m^2), intravenously (IV), once weekly for 4 weeks. Participants who achieved minor response (MR), partial response (PR), or complete response (CR) after the first cycle received a second cycle of treatment for a maximum of 2 cycles.
- Rituximab + Interferon (IFN): Participants received rituximab 375 mg/m^2, IV, once weekly for 4 weeks. Participants also received IFN-alpha2a (IFN-α2a), 3 million international units per day (MIU/day), subcutaneously (SC), during Week 1, and 4.5 MIU/day, SC, 6 days per week during Weeks 2 through 5. IFN-α2a was not administered on days of rituximab administration. Participants who achieved MR, PR, or CR during the first cycle received a second cycle of treatment for a maximum of 2 cycles.
Period: Overall Study
Arm/Group | Rituximab Monotherapy | Rituximab + Interferon (IFN)
Started | 156 | 157
Entering Cycle 2 | 120 | 124
Completed | 113 | 120
Not Completed | 43 | 37
Not completed — Stable disease (SD) | 22 | 16
Not completed — Progressive disease (PD) | 8 | 10
Not completed — Adverse Event | 3 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Other | 2 | 0
Not completed — Other malignancy | 1 | 0
Not completed — Pathology review | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — New cancer | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants.
Groups:
- Rituximab Monotherapy: Participants rituximab received 375 mg/m^2, IV, once weekly for 4 weeks. Participants who achieved MR, PR, or CR after the first cycle received a second cycle of treatment for a maximum of 2 cycles.
- Rituximab + IFN: Participants received rituximab 375 mg/m^2, IV, once weekly for 4 weeks. Participants also received IFN-α2a 3 MIU/day, SC, during Week 1, and 4.5 MIU/day, SC, 6 days per week during Weeks 2 through 5. IFN-α2a was not administered on days of rituximab administration. Participants who achieved MR, PR, or CR during the first cycle received a second cycle of treatment for a maximum of 2 cycles.
- Total: Total of all reporting groups
Arm/Group | Rituximab Monotherapy | Rituximab + IFN | Total
Number analyzed (Participants) | 156 | 157 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (11.6) | 57.2 (10.8) | 58.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 82 | 160
  Male | 78 | 75 | 153

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure - Percentage of Participants With an Event
Description: Treatment failure was defined as an event of any of the following: progressive disease while receiving study treatment, death due to any cause, or the initiation of another type of treatment due to stable disease, progressive disease or relapse, or intolerance to study treatment.
Time Frame: Baseline (BL), Week 10 and 16, and Months 6, 12, 18, 24, 30, and 42 of the follow-up period
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 156 | 157
percentage of participants | 68 | 67

2. Primary Outcome: Treatment Failure - Time to Event
Description: The median time, in months, between randomization and treatment failure event determined using Kaplan-Meier estimates.
Time Frame: BL, Week 10 and 16, and Months 6, 12, 18, 24, 30, and 42 of the follow-up period
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 156 | 157
months | 21.5 [13.6 to 26.5] | 28.0 [20.7 to 41.0]
Statistical Analysis 1: Comparison: Rituximab Monotherapy vs Rituximab + IFN; Test type: Superiority or Other; p = 0.3023, Log Rank

3. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR), Unconfirmed CR (CRu), or Partial Response (PR)
Description: CR was defined as the complete disappearance of all previously detectable disease signs; the absence of palpable lymph nodes greater than (>) 1 centimeter (cm) or nodes >1.5 cm observed in computerized axial tomography (CAT) scan; and negative bone marrow pathology, if initially positive. CRu was defined as CR, except that bone marrow results were indeterminate. PR was defined as a decrease of greater than or equal to (≥) 50 percent (%) compared with the BL value in the sum of the products of the two largest perpendicular diameters in all measurable and evaluable lesions; and a ≥50% reduction of the size from BL if hepato-splenomegaly was present.
Time Frame: Weeks 10 and 16
Population: ITT population; number (n) equals (=) number of participants assessed for the specified parameter at a given visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 156 | 157
percentage of participants
  Week 10, Cycle 1 (n=156,157) | 54 [46 to 62] | 59 [51 to 67]
  Week 16, Cycle 2 (n=123,124) | 74 [65 to 81] | 82 [74 to 89]
Statistical Analysis 1: Comparison: Rituximab Monotherapy vs Rituximab + IFN; Week 10, Cycle 1; Test type: Superiority or Other; p = 0.3362, Chi-squared
Statistical Analysis 2: Comparison: Rituximab Monotherapy vs Rituximab + IFN; Week 16, Cycle 2; Test type: Superiority or Other; p = 0.1157, Chi-squared

4. Secondary Outcome: Percentage of Participants Achieving CR or CRu
Description: CR was defined as the complete disappearance of all previously detectable disease signs; the absence of palpable lymph nodes >1 cm or nodes >1.5 cm observed in CATscan; and negative bone marrow pathology, if initially positive. CRu was defined as CR, except that bone marrow results were indeterminate.
Time Frame: Weeks 10 and 16
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 156 | 157
percentage of participants
  Week 10, Cycle 1 (n=156,157) | 8 [5 to 14] | 9 [5 to 15]
  Week 16, Cycle 2 (n=123,124) | 24 [17 to 33] | 41 [32 to 50]
Statistical Analysis 1: Comparison: Rituximab Monotherapy vs Rituximab + IFN; Week 10, Cycle 1; Test type: Superiority or Other; p = 0.8540, Chi-squared
Statistical Analysis 2: Comparison: Rituximab Monotherapy vs Rituximab + IFN; Week 16, Cycle 2; Test type: Superiority or Other; p = 0.0051, Chi-squared

5. Secondary Outcome: Duration of Response - Percentage of Participants With an Event
Description: Response duration was defined as the period between the date for first observation of CR, CRu or PR and the date of progressive disease (PD), censored observation or death of any cause. Response duration was also assessed for response defined as CR only. Response duration was calculated among responders (CR+CRu+PR) with cutoffs for follow-up applied.
Time Frame: BL, Week 10 and 16, and Months 6, 12, 18, 24, 30, and 42 of the follow-up period
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 102 | 113
percentage of participants
  CR, CRu, and PR (n=102,113) | 63 | 65
  CR and CRu only (n=62,73) | 44 | 53
  CR only (n=50,62) | 38 | 48

6. Secondary Outcome: Duration of Response
Description: The median time, in months, from the date of the first observation of CR, CRu, or PR and the date of progressive disease (PD), censored observation, or death due to any cause. PD was defined as an increase of >50% compared to BL in the sum of the product of the two largest perpendicular parameters of measurable lymphoma, or the occurrence of new lesions. One month=30.4 days. Response duration was calculated amongst responders (CR+CRu+PR) with cutoffs for follow-up applied.
Time Frame: BL, Week 10 and 16, and Months 6, 12, 18, 24, 30, and 42 of the follow-up period
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit. Only participants with a response (CR+CRu+PR, CR+CRu, or CR only) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 156 | 157
months
  CR+CRu+PR (n=102,113) | 22.0 [15.9 to 32.3] | 30.0 [20.1 to 39.8]
  CR+CRu only (n=62,73) | NA [23.0 to NA] — The median and upper limit of the 95% confidence interval (CI) were not estimable due to censoring. | 44.4 [33.0 to NA] — The upper limit of the 95% CI was not estimable due to censoring.
  CR only (n=50,62) | 59.5 [23.1 to NA] — The upper limit of the 95% CI was not estimable due to censoring. | 50.7 [26.7 to NA] — The upper limit of the 95% CI was not estimable due to censoring.
Statistical Analysis 1: Comparison: Rituximab Monotherapy vs Rituximab + IFN; CR+CRu+PR; Test type: Superiority or Other; p = 0.7840, Log Rank; Stratification by previous treatment for lymphoma (yes or no)
Statistical Analysis 2: Comparison: Rituximab Monotherapy vs Rituximab + IFN; CR+CRu; Test type: Superiority or Other; p = 0.4419, Log Rank; Stratification by previous treatment for lymphoma (yes or no)
Statistical Analysis 3: Comparison: Rituximab Monotherapy vs Rituximab + IFN; CR only; Test type: Superiority or Other; p = 0.5942, Log Rank; Stratification by previous treatment for lymphoma (yes or no)

7. Secondary Outcome: Disease Progression - Percentage of Participants With an Event
Description: A disease progression event was defined as tumor progression or death due to any cause (or a censored observation).
Time Frame: BL, Week 10 and 16, and Months 6, 12, 18, 24, 30, and 42 of the follow-up period
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 156 | 157
percentage of participants | 60 | 62

8. Secondary Outcome: Time to Disease Progression
Description: The median time, in months, from randomization to disease progression event assessed using Kaplan-Meier estimates. One month=30.4 days
Time Frame: BL, Week 10 and 16, and Months 6, 12, 18, 24, 30, and 42 of the follow-up period
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 156 | 157
months | 25.0 [18.7 to 39.8] | 32.0 [21.7 to 40.3]
Statistical Analysis 1: Comparison: Rituximab Monotherapy vs Rituximab + IFN; Test type: Superiority or Other; p = 0.8946, Log Rank; Stratified by previous treatment for lymphoma (yes or no)

9. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: An overall survival event was defined as death due to any cause.
Time Frame: BL, Week 10 and 16, and Months 6, 12, 18, 24, 30, and 42 of the follow-up period
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 156 | 157
percentage of participants | 13 | 11

10. Secondary Outcome: Overall Survival
Description: The median time, in months, from randomization to OS event assessed using Kaplan-Meier estimates. One month=30.4 days
Time Frame: BL, Week 10 and 16, and Months 6, 12, 18, 24, 30, and 42 of the follow-up period
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Number analyzed (Participants) | 156 | 157
months | NA [3.6 to 98.9] — Median OS had not been reached at time of analysis. | NA [3.4 to 97.8] — Median OS had not been reached at time of analysis.
Statistical Analysis 1: Comparison: Rituximab Monotherapy vs Rituximab + IFN; Test type: Superiority or Other; p = 0.4963, Log Rank; Stratified by previous treatment for lymphoma (yes or no)

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events (AEs) from BL, Weeks 1 through 16, and Months 6, 12, 18, 24, 30, and 42 of the follow-up period.
Description: Nonserious AEs presented in this record include all AEs reported during the study, not just nonserious events. Additionally, AE information is presented by system organ class (SOC) as AE data by preferred term were not available within the specified parameters (that is, with 5% threshold).
Arm/Group | Rituximab Monotherapy | Rituximab + IFN
Serious Adverse Events (participants affected / at risk) | 13/156 | 34/157
Other Adverse Events (participants affected / at risk) | 138/156 | 155/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Monotherapy (N=156) | Rituximab + IFN (N=157)
General disorders and administration site conditions (ASC) (General disorders) | 2 | 9
Gastrointestinal disorders (Gastrointestinal disorders) | 4 | 6
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 | 6
Respiratory, thoracic and mediastinal (T&M) disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Infections and infestations (Infections and infestations) | 3 | 5
Nervous system disorders (Nervous system disorders) | 1 | 4
Musculoskeletal and connective tissue (CT) disorders (Musculoskeletal and connective tissue disorders) | 1 | 2
Immune system disorders (Immune system disorders) | 1 | 1
Investigations (Investigations) | 0 | 1
Cardiac disorders (Cardiac disorders) | 1 | 2
Injury, poisoning and procedural complications (PC) (Injury, poisoning and procedural complications) | 0 | 3
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 | 2
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 1
Psychiatric disorders (Psychiatric disorders) | 0 | 1
Vascular disorders (Vascular disorders) | 1 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 | 1
Eye disorders (Eye disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (including cysts) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Monotherapy (N=156) | Rituximab + IFN (N=157)
General disorders and ASC (General disorders) | 70 | 141
Gastrointestinal disorders (Gastrointestinal disorders) | 48 | 101
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 35 | 81
Nervous system disorders (Nervous system disorders) | 22 | 82
Infections and infestations (Infections and infestations) | 38 | 58
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 29 | 65
Respiratory, T&M disorders (Respiratory, thoracic and mediastinal disorders) | 37 | 32
Psychiatric disorders (Psychiatric disorders) | 11 | 38
Vascular disorders (Vascular disorders) | 21 | 16
Immune system disorders (Immune system disorders) | 15 | 18
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 6 | 20
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 | 23
Investigations (Investigations) | 6 | 14
Eye disorders (Eye disorders) | 3 | 16
Cardiac disorders (Cardiac disorders) | 7 | 9
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 | 8
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 11
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 | 7
Renal and urinary disorders (Renal and urinary disorders) | 5 | 2
Neoplasms benign, malignant and unspecified (including cysts) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Surgical and medical procedures (Surgical and medical procedures) | 1 | 0

LIMITATIONS AND CAVEATS:
Nonserious AEs presented in this record include all AEs reported during the study, not just nonserious events, and information is presented by SOC as AE data by preferred term were not available within specified parameters (with 5% threshold).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.